CLINICAL TRIAL: NCT01925027
Title: Efficacy and Safety of Nano+ Polymer-free Sirolimus-Eluting Stent in the Treatment of Patients With De Novo Lesion: A Optical Coherent Tomography Prospective, Multicenter Study
Brief Title: Efficacy and Safety of Nano+ Polymer-free Sirolimus-Eluting Stent: A Optical Coherent Tomography Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120025
Record Dates: First submitted 2013-08-04; First posted 2013-08-19 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Nano+ DES; OCT; Neointimal hyperplasia; DAPT; 3 month
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NANO+ DES (Experimental): The Nano+ Polymer-free Sirolimus-Eluting Coronary Stent System is device/drug combination products consisting of a drug-coated stent and a balloon expandable delivery system. The stent is coated with a formulation containing rapamycin, the active ingredient, adhered to 316L stainless bare stent scaffold with submicron micropores, and is approved by State Food and Drug Administration of China in 2011(No. 3460037).
  Interventions: Device: Nano+ DES

INTERVENTIONS:
Device: Nano+ DES — All patients will be treated with the NanoTM Polymer-free Sirolimus Coronary Stent System. All patients will undergo angiographic (QCA) investigation at baseline (pre- and post-procedure) and at 3 months follow-up. All patients will undergo OCT investigation at 3 months follow-up. All patients will be evaluated clinically at 3, 4, 5 months (for patients with 6 months OCT follow-up evaluation will be at 8 months) and at 1 and 2 years.
  Other Names: NANO+ Polymer-free Sirolimus-Eluting Stent

SUMMARY:
Our hypothesis is to test that 1) The safety and efficacy of Nano+ DES in patients with de novo lesions; 2) A low neointimal hyperplasia after Nano+ DES implantation due to its effective and sufficient antiproliferative drug; 3) A very high coverage and an improved early arterial healing after Nano+ DES implantation due to polymer-free; 4) The safety of clopidogrel treatment discontinuation at 3 months when OCT results are defined as optimal.

DETAILED DESCRIPTION:
Eligibility criteria:

* 18 to 85 years.
* Evidence of myocardial ischemia without raised troponin (e.g. stable or unstable angina, silent ischemia demonstrated by positive territorial functional study).
* The patient has a planned intervention of up to two de novo lesions in different epicardial vessels
* Lesion(s) must have a visually estimated diameter stenosis of ≥50% and <100%.
* Lesion length must be <18mm
* RVD must be between 2.5-4.0 mm
* Written informed consent.
* The patient and the patient's physician agree to the follow-up visits including angiographic follow-up and OCT assessment at 3 months.

Design details and outcomes This is a prospective, multicentre, single arm, open- label study, which will enroll a total of 45 patients in 5 European investigational sites. All patients will be treated with the Nano+ Polymer-free Sirolimus Coronary Stent System. All patients will undergo angiographic (QCA) investigation at baseline (pre- and post-procedure) and at 3 months follow-up. All patients will undergo OCT investigation at 3 months follow-up. OCT investigation will be performed at 6 months follow-up in those patients where the OCT criteria (coverage and stent apposition) were not met at 3 months OCT. Off-line OCT and angiographic data analysis will be undertaken by an independent core laboratory (Cardialysis BV, Rotterdam, The Netherlands) blinded to clinical and procedural characteristics of the patients and according to pre-set Standard Operating Procedures. All patients will be evaluated clinically at 3, 4, 5 months (for patients with 6 months OCT follow-up evaluation will be at 8 months) and at 1 and 2 years. Clinical data will be adjudicated by an independent Clinical Event Committee. An independent Data Safety and Monitoring Board (DSMB) will monitor the individual and collective safety of the patients in the study on an ongoing basis. This is a hypothesis generating study, because no evidence about the expected magnitude of the effect is available at present. Data generated from this study will be compared (historical control) against historical figures of other drug eluting stents available at Cardialysis, for published data.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years.
* Evidence of myocardial ischemia without raised troponin (e.g. stable or unstable angina, silent ischemia demonstrated by positive territorial functional study).
* The patient has a planned intervention of up to two de novo lesions in different epicardial vessels
* Lesion(s) must have a visually estimated diameter stenosis of ≥50% and <100%.
* Lesion length must be <18mm
* RVD must be between 2.5-4.0 mm
* Written informed consent.
* The patient and the patient's physician agree to the follow-up visits including angiographic follow-up and OCT assessment at 3 months.

Exclusion Criteria:

* Evidence of ongoing acute myocardial infarction in ECG prior to procedure.
* LVEF <30%.
* Platelet count <100,000 cells/mm3 or >700,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis).
* Known renal insufficiency (e.g., eGFR <60 ml/kg/m2 or serum creatinine level of >2.5 mg/dL, or subject on dialysis).
* History of bleeding diathesis or coagulopathy.
* The patient is a recipient of a heart transplant.
* Known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel prasugrel, ticagrelor and ticlopidine), sirolimus or stainless steel.
* Other medical illness (e.g. cancer, stroke with neurological deficiency) or known history of substance abuse (alcohol, cocaine, heroin etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy
* Participating in other drugs or medical devices clinical trials, prior to reaching the primary endpoint.
* Pregnant or breastfeeding woman or woman in fertile period not taking adequate contraceptives

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
In-stent neointimal hyperplasia volume obstruction (%) | 3-month
  For those patients that did not achieve the optimal/ successful OCT criteria at 3 months an additional OCT investigation will be planned at 6 months follow-up where these same endpoints will be assessed.

SECONDARY OUTCOMES:
Neointimal hyperplasia area/volume | 3-month
Mean/Minimal Stent diameter/area/volume | 3-month
Mean/Minimal Lumen diameter/area/volume | 3-month
Mean/maximal thickness of the struts coverage | 3-month
Percentage of covered struts | 3-month
Incomplete strut apposition | 3-month

OTHER OUTCOMES:
MLD and %DS | 3-month
  All measurements will be made of the in-stent, in-segment, proximal and distal stent margins.
Late Lumen Loss | 3-month
  The difference between the minimum lumen diameter (MLD) post procedure and the MLD at 3 month follow-up.
Binary Restenosis (DS ≥50%) | 3-month
Acute success | 3 month
  Acute success will be classified according to the following definitions:
  1. Device success: < 30% residual stenosis (by on-line QCA)
  2. Procedure success: The attainment of < 30% residual stenosis by QCA AND either a TIMI flow 3 or a consistent TIMI flow 2 before and after the procedure, using any percutaneous method without the occurrence of MACE during the hospital stay. These measurements will be made by the independent angiographic core laboratory. If the core laboratory is unable to assess the % residual stenosis, the investigator's assessment as recorded in the CRF will be used for the statistical analysis.
Device-oriented Composite Endpoints and its individual component | up to 2 years
  Device-oriented Composite Endpoint (DoCE) is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization
Stent thrombosis | up to 2 years
  According to the ARC definitions

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, PhD, Study Chair — Erasmus Medical Center; Run-Lin Gao, MD, Principal Investigator — Fu Wai Hospital, Beijing, China; Bo Xu, MSc, Principal Investigator — Fu Wai Hospital, Beijing, China; Yao-Jun Zhang, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (5):
- Belgium (2):
  - UZ Virga Jesse Ziekenhuis, Hasselt
  - CHU Sart Tillman, Liège
- Netherlands (3):
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Erasmus Medical Centre, Rotterdam